CLINICAL TRIAL: NCT03824405
Title: A Randomized, Double-Blind, Vehicle-Controlled Study of the Safety, Tolerability and Efficacy of BTX 1204 in Patients With Moderate Atopic Dermatitis
Brief Title: Study of the Safety, Tolerability and Efficacy of BTX 1204 in Patients With Moderate Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Botanix Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTX.2018.003
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-09

CONDITIONS: Atopic Dermatitis
Keywords: CBD; Synthetic CBD; Cannabidiol
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BTX 1204 (Active Comparator): BTX 1204 twice daily
  Interventions: Drug: BTX 1204
- Vehicle (Placebo Comparator): Vehicle twice daily
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: BTX 1204 — BTX 1204 liquid formulation
  Arms: BTX 1204
Drug: Vehicle — Vehicle liquid formulation
  Arms: Vehicle

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, Phase 2 study in subjects with moderate AD.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled, Phase 2 study in subjects with moderate AD. Eligible subjects will be enrolled and randomized to treatment with BTX 1204 or Vehicle for 84 days. Approximately two hundred (200) subjects will be enrolled. Subjects will receive BID application of study drug for 84 days with a final application on the evening of Day 84 for a total of 168 doses.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is of either gender between 12 and 70 years of age, inclusive.
2. Subject (or parent/legal guardian) has the ability and willingness to sign a written informed consent.
3. Subject has a diagnosis of chronic (≥1 year), stable atopic dermatitis (AD)
4. Subject has ≥ 5% and ≤ 30% body surface area (BSA) of AD involvement excluding the scalp and groin.
5. Subject has an Investigator's Global Assessment (IGA) score of moderate (3) atopic dermatitis on the 5-point IGA (0-4) scale.
6. For selected photography sites, subject has a target lesion of 25 to 200 cm2 in surface area on the trunk, upper extremities or lower extremities with a Baseline Signs of AD score of ≥ 6 and ≤ 12.
7. Subject is in good general health without clinically significant hematological, cardiac, respiratory, renal, endocrine, gastrointestinal, psychiatric, hepatic, or malignant disease, as determined by the investigator.
8. Subject has suitable venous access for blood sampling.
9. Subject is able and willing to complete the study and to comply with all study instructions and attend the necessary visits.
10. Male subjects and their partners must agree and commit to use a barrier method of contraception throughout the study and for 90 days after last study drug application.
11. A negative urine pregnancy test result for all Women of child bearing potential (WOCBP) at the Screening Visit and Baseline Visit.
12. Sexually active women must agree to use the following throughout the study and for 30 days after last study drug application. WOCBP who are not sexually active at Baseline and become sexually active must identify a plan for contraception.

    1. One of these highly effective contraception methods Intrauterine device (IUD); hormonal (injections, implants, transdermal patch, vaginal ring); tubal ligation; partner vasectomy, OR
    2. Oral contraceptives WITH a barrier method (listed below), OR
    3. Two barrier forms of contraception (listed below) Male or female condom; diaphragm; cervical cap; contraceptive sponge.
13. Males subjects must refrain from sperm donation during the study treatment period and until 90 days after last study drug application.

Exclusion Criteria:

1. Female subject who is breast feeding, pregnant, or planning to become pregnant.
2. Subject who has an IGA score of 2 (mild) or 4 (severe).
3. Subject with history of known or suspected intolerance to the drug product excipients.
4. Subject has any clinically significant active infection in the investigator's opinion. This includes active impetigo at any AD lesion.
5. Subject has known Hepatitis-B, Hepatitis-C, or HIV infection.
6. Subject has excessive body or facial hair that would interfere with the evaluation of safety or with the diagnosis or assessment of AD.
7. Subject has sunburns, unevenness in skin tones, tattoos, scars, excessive hair, freckles, birthmarks, moles, or other skin damage or abnormality that would result in the inability to evaluate the AD lesions.
8. Subject has clinically significant or severe allergies that in the investigator's opinion would interfere with participation in the study.
9. Subject has known intolerability to topical treatments e.g., reports excessive burning/stinging or pain with use of topical treatments.
10. Subject has an active or potentially recurring skin conditions(s) other than AD that in the investigator's opinion would interfere with participation in the study.
11. Subject has unstable AD consistent with a requirement for high-potency corticosteroids.
12. Subject has used dupilumab (Dupixent) within 12 weeks prior to the Baseline Visit.
13. Subject has used any biologic therapy, other than dupilumab, within 28 days prior to the Baseline Visit.
14. Subject has used systemic (oral, IV or IM) corticosteroids within 28 days prior to the Baseline Visit. Intra-articular injection for arthroses allowed.
15. Subject has used topical anti-pruritics (e.g., PDE4 inhibitors) within 28 days prior to the Baseline Visit.
16. If subject is taking oral antihistamines, subject has not been on a stable dose of oral antihistamines within 28 days prior to the Baseline visit.
17. Subject has used phototherapy, tanning beds, or any other artificial light device within 28 days prior to the Baseline Visit.
18. Subject has used topical corticosteroids within 14 days prior to the Baseline Visit.
19. Subject has used topical calcineurin inhibitors within 14 days prior to the Baseline Visit.
20. Subjects has used barrier creams (e.g., Mimyx, Atopiclair), within 7 days prior to the Baseline Visit.
21. Subject has an underlying disease that requires the use of interfering topical or systemic therapy.
22. Subject has other dermatological conditions that require the use of interfering topical or systemic therapy or that might interfere with study assessments such as, but not limited to, acne or rosacea.
23. Subject has a clinically relevant history or currently suffering from any disease or condition that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk or interfere with the subject's participation in the study. Subjects with other dermatologic conditions, including genetic syndromes that have an eczematous dermatitis as a component of the disease (e.g., Netherton's) are excluded.
24. Subject has a clinically relevant history of or current evidence of abuse of alcohol or other drugs.
25. Subject is currently using any medication that, in the opinion of the investigator, may affect the evaluation of the study product or place the subject at undue risk.
26. Subject has participated in another investigational drug or device research study within 30 days of the Screening Visit or five half-lives of the drug, whichever is longer.
27. Any other reason that would make the subject, in the opinion of the Investigator or sponsor, unsuitable for the study.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Robinson, CRNP, Study Director — Head of Development, Botanix Pharmaceuticals
Locations (31):
- United States (19):
  - Applied Research Center of Arkansas Inc., Little Rock, Arkansas
  - T. Joseph Raoff MD Inc. / Encino Research Center, Encino, California
  - Center for Dermatology Clinical Research, Fremont, California
  - Dermatology Specialist Inc. - Murrieta, Murrieta, California
  - Rady Childern's Hospital - San Diego, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Precision Clinical Research, Davie, Florida
  - Troy Sullivan, North Miami Beach, Florida
  - DS Research, Louisville, Kentucky
  - Delright Research, New Orleans, Louisiana
  - Medisearch Clinical Trails, Saint Joseph, Missouri
  - Washington Univerisy in St. Louis, St Louis, Missouri
  - JDR Dermatology Research LLC, Las Vegas, Nevada
  - The Acne Treatment and Research Center, Morristown, New Jersey
  - Aventiv Research Inc - Dublin, Dublin, Ohio
  - Greenville Dermatology, LLC, Greenville, South Carolina
  - Dermresearch Inc, Austin, Texas
  - J&S Studies Inc., College Station, Texas
  - The Center for Skin Research at Suzanne Bruce & Associates Dermatology, Houston, Texas
- Australia (9):
  - CMAX Clincial Research, Adelaide
  - BurwoodDermatology, Burwood
  - Sinclair Dermatology, East Melbourne
  - North Eastern Health Specialists, Hectorville
  - Premier Specialists PTY LTD, Kogarah
  - St George Dermatology & Skin Cancer Center, Kogarah
  - Captain Stirling Medical Centre, Nedlands
  - The Skin Hospital, Westmead
  - Veracity Clinical Research, Woolloongabba
- New Zealand (3):
  - Optimal Clinical Trials, Auckland
  - Clinical Trials New Zealand LTD, Hamilton
  - P3 Research, Wellington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BTX 1204 | Vehicle
Started | 100 | 100
Completed | 65 | 55
Not Completed | 35 | 45

BASELINE CHARACTERISTICS:
Population: Intent-to-treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | BTX 1204 | Vehicle | Total
Number analyzed (Participants) | 99 | 95 | 194
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20 | 15 | 35
  Between 18 and 65 years | 77 | 76 | 153
  >=65 years | 2 | 4 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 54 | 116
  Male | 37 | 41 | 78
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 11 | 20
  Not Hispanic or Latino | 90 | 84 | 174
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 18 | 17 | 35
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 14 | 18 | 32
  White | 53 | 55 | 108
  More than one race | 11 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0
Investigator Global Assessment [Count of Participants; unit: Participants]
  0 - Clear | 0 | 0 | 0
  1 - Almost Clear | 0 | 0 | 0
  2 - Mild | 0 | 0 | 0
  3 - Moderate | 99 | 95 | 194
  4 - Severe | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Investigator's Global Assessment (IGA)
Description: Investigator's Global Assessment (IGA) success defined as an IGA score of "Clear" (0) or "Almost Clear" (1) with at least a 2-grade improvement
Time Frame: Day 85
Population: ITT Summary of Subjects Excluded From Analyses (Randomized Subjects) BTX 1204 4% BID (N=100) Vehicle BID (N=100)
  Number of Subjects Excluded from the ITT Population, n (%) BTX 1204 4% BID 1 (1.0) Vehicle BID 5 (5.0)
  Reason for Exclusion from the ITT Population, n (%) Not At Least One Post-Baseline Efficacy Assessment BTX 1204 4% BID 1 (1.0) Vehicle BID 5 (5.0)
Measure: Count of Participants; unit: Participants
Arm/Group | BTX 1204 | Vehicle
Number analyzed (Participants) | 99 | 95
Participants
  Success | 12 | 18
  Failure | 87 | 77

ADVERSE EVENTS:
Time Frame: 85 days
Description: Summary of Subjects Excluded From Analyses (Randomized Subjects) BTX 1204 4% BID (N=100) Vehicle BID (N=100)
  Number of Subjects Excluded from the Safety Population, n (%) BTX 1204 4% BID 1 (1.0) Vehicle BID 2 (2.0)
  Reason for Exclusion from the Safety Population, n (%) No Post-Baseline Safety Assessment BTX 1204 4% BID 1 (1.0) Vehicle BID 2 (2.0)
Arm/Group | BTX 1204 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/98
Serious Adverse Events (participants affected / at risk) | 2/99 | 0/98
Other Adverse Events (participants affected / at risk) | 37/99 | 25/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BTX 1204 (N=99) | Vehicle (N=98)
Post-procedural complication (General disorders) | 1 | 0 — Outcome: Recovered/resolved Severity: Severe Causality: Unrelated Study Drug Action Taken: None
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — Outcome: Recovered/resolved Causality: Unrelated Study Drug Action Taken: Not Applicable
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BTX 1204 (N=99) | Vehicle (N=98)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 15
Erythema (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Nasopharyngitis (Skin and subcutaneous tissue disorders) | 6 | 1
Application Site Pain (Skin and subcutaneous tissue disorders) | 4 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 3
Application Site Reaction (Skin and subcutaneous tissue disorders) | 3 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As Study is a Multi-centre Study, no Publication of the Study results may be made until Publication of the results of the Multi-centre study or 2 years after Study Completion, whichever is sooner.

DOCUMENTS (2):
  • Study Protocol (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/05/NCT03824405/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT03824405/SAP_001.pdf